CLINICAL TRIAL: NCT03082820
Title: Evaluation of Pain-related Evoked Potentials (PREP) for the Objectivization of Neuropathic Pain
Brief Title: Pain-related Evoked Potentials in Unilateral Peripheral Nerve Injuries
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof. Dr. med., Ruhr University of Bochum
Other Study IDs: PREP2015
Record Dates: First submitted 2017-03-06; First posted 2017-03-17 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Peripheral Nerve Injuries
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Nerve Conduction Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Pain-related evoked potentials (PREP), Quantitative Sensory Testing (QST) and nerve conduction studies (NCS) were performed with patients with peripheral nerve injury.
  Interventions: Diagnostic Test: Pain-related evoked potentials (PREP); Diagnostic Test: Quantitative Sensory Testing (QST); Diagnostic Test: Nerve conduction studies (NCS)
- Controls: Pain-related evoked potentials (PREP) and Quantitative Sensory Testing (QST) were performed with healthy adults.
  Interventions: Diagnostic Test: Pain-related evoked potentials (PREP); Diagnostic Test: Quantitative Sensory Testing (QST)

INTERVENTIONS:
Diagnostic Test: Pain-related evoked potentials (PREP) — PREP were performed bilaterally with a concentric surface electrode at twice the individual pain threshold.
Diagnostic Test: Quantitative Sensory Testing (QST) — QST was performed bilaterally following the protocol of the German Network on Neuropathic Pain.
Diagnostic Test: Nerve conduction studies (NCS) — NCS were performed with patients only.
  Groups: Patients

SUMMARY:
The study examines pain-related evoked potentials (PREP) in patients with peripheral nerve injuries. Since previous studies found altered latencies and amplitudes of PREP in generalized polyneuropathies, e. g. HIV-polyneuropathy and fibromyalgia, this study investigates if these alterations are detectable in unilateral peripheral nerve injuries as well.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral Nerve Injury

Exclusion Criteria:

* Polyneuropathy
* Contralateral peripheral nerve injury
* Severe psychiatric disorders
* Disorders affecting central nervous system

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with PNI treated in the university hospital Bergmannsheil Bochum, Bochum, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2015-02-03; Primary Completion 2016-11-05 (Actual); Study Completion 2016-11-05 (Actual)

PRIMARY OUTCOMES:
N1-latency | 1 day
  N1-latency of pain-related evoked potentials in ms

SECONDARY OUTCOMES:
N1P1-amplitude | 1 day
  Amplitude of pain-related evoked potentials in µV

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof. Dr. med., Study Director — University Hospital Bergmannsheil Bochum

IPD SHARING:
Plan to Share IPD: No